CLINICAL TRIAL: NCT06576986
Title: Effect of Synbiotic Supplementation on the Prevention of Mucositis in Cancer Patients Undergoing Chemotherapy: Randomized, Double-masked, Parallel, Single-center Clinical Trial
Brief Title: Effect of Synbiotic Supplementation on the Prevention of Mucositis in Cancer Patients Undergoing Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Principal Investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 30177920200005149
Record Dates: First submitted 2024-05-11; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Colo-rectal Cancer
Keywords: colorectal cancer; symbiotic; Mucositis; diarrhea; chemotherapy
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Mucositis; Diarrhea | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Capecitabine alone control (Placebo Comparator): n the Control Group, patients received Maltodextrin as supplementation
  Interventions: Dietary Supplement: Maltodextrin
- Capecitabine alone synbiotic (Experimental): In the Intervention Group, patients received the symbiotic Simbioflora as supplementation.
  Interventions: Dietary Supplement: Symbiotic
- Capecitabine associated with control Oxaliplatin (Placebo Comparator): n the Control Group, patients received Maltodextrin as supplementation
  Interventions: Dietary Supplement: Maltodextrin
- Capecitabine associated with synbiotic Oxaliplatin (Experimental): In the Intervention Group, patients received the symbiotic Simbioflora as supplementation.
  Interventions: Dietary Supplement: Symbiotic

INTERVENTIONS:
Dietary Supplement: Symbiotic — The synbiotic used will be Simbioflora® (commercial preparation containing 5.5g of FOS added with four species of probiotic, Lactobacillus paracasei LPC-31; Lactobacillus rhamnosus HN001; Lactobacillus acidophilus NCFM; Bifidobacterium lactis HN019, at a concentration of 109 UFC per strain) supplied by Farmoquímica S.A. Supplementation will be administered orally, twice a day, before lunch and dinner, for ten days before chemotherapy treatment. Patients will be guided by researchers on dilution (100 mL of filtered water) and the correct purchase of the modules. Consumption control will be carried out daily, via telephone contact.
  Other Names: Simbioflora
  Arms: Capecitabine alone synbiotic; Capecitabine associated with synbiotic Oxaliplatin
Dietary Supplement: Maltodextrin — Maltodextrin, used as control, will be purchased from the company PRODIET® under the trade name Carboch®. Supplementation will be administered orally, twice a day, before lunch and dinner, for ten days before chemotherapy treatment. Patients will be guided by researchers on dilution (100 mL of filtered water) and the correct purchase of the modules. Consumption control will be carried out daily, via telephone contact.
  Arms: Capecitabine alone control; Capecitabine associated with control Oxaliplatin

SUMMARY:
Introduction: In the 2023-2025 period, colorectal cancer (CRC) will be the third most common type of cancer in Brazil. The most commonly used therapeutic approaches are chemotherapy (QTx) and radiotherapy (RTx). QTx agents, such as capecitabine, affect both malignant cells and normal cells such as gastrointestinal, capillary and immune cells. Cellular damage in the gastrointestinal tract (GIT) results in various symptoms, such as mucositis and diarrhea. Diarrhea is linked to mucosal damage and can result in dehydration, malnutrition and hospitalization, leading to cardiovascular complications and death. Mucositis is inflammation that affects the GIT. This condition makes treatment difficult, leading to reductions, delays or interruption of QTx. These scenarios harm the patient's prognosis and quality of life, resulting in high costs for symptom control, nutritional assistance, management of secondary infections and hospitalization. The Mucositis Study Group (MASCC/ISOO) guidelines recommend the use of probiotics as a preventive measure against diarrhea in cancer patients undergoing QTx and/or RTx. However, the safety of using probiotics in immunosuppressed patients is still controversial and hypotheses are based on epidemiological and experimental studies. This makes it necessary to evaluate whether supplementation with pro- or synbiotics before chemotherapy would have the same beneficial results. Objective: To evaluate the effect of synbiotic supplementation on the prevention, incidence and severity of mucositis in cancer patients undergoing QTx. Method: This is a single-center parallel double-masked randomized clinical trial to be carried out at the Borges da Costa/UFMG Outpatient Clinic at Hospital das Clínicas in Belo Horizonte - Minas Gerais (HC-BH/MG). The inclusion criteria are patients diagnosed with CRC eligible for first-line treatment with Capecitabine, aged ≥ 18 years, both sexes, signed the informed consent form. The study was approved by CEP-UFMG. Expected results: It is expected that supplementation with synbiotics in the pre-QTx period will promote modulation of the microbiota and strengthening of the intestinal barrier, resulting in a lower incidence and severity of mucositis and diarrhea, improving the quality of life of these patients.

DETAILED DESCRIPTION:
Introduction: In the triennium 2023-2025, colorectal cancer (CRC) will be the third most common type of cancer in Brazil. The most used therapeutic approaches are chemotherapy (QTx) and radiotherapy (RTx). Chemotherapeutic agents, such as capecitabine, affect both malignant cells and normal cells such as gastrointestinal, capillary, and immune cells. Cellular damage in the gastrointestinal tract (GIT) results in various symptoms, such as mucositis and diarrhea. Diarrhea is linked to mucosal injury and can lead to dehydration, malnutrition, hospitalization, cardiovascular complications, and death. Mucositis, on the other hand, is inflammation that affects the GIT. This condition hinders treatment, leading to reductions, delays, or interruption of QTx. These scenarios impair the prognosis and quality of life of the patient, resulting in high costs for symptom control, nutritional support, management of secondary infections, and hospitalization. The Mucositis Study Group guidelines (MASCC/ISOO) recommend the use of probiotics as a preventive measure against diarrhea in cancer patients undergoing QTx and/or RTx. However, the safety of probiotic use in immunosuppressed patients is still controversial, and hypotheses are based on epidemiological and experimental studies. Therefore, it is necessary to evaluate whether supplementation with probiotics or symbiotics before chemotherapy would have the same beneficial results. Objective: The general objective of this study is to evaluate if symbiotic supplementation can reduce the incidence and severity of oral mucositis in cancer patients undergoing chemotherapy. Specific objectives include assessing the tolerability of supplementation, analyzing clinical and laboratory parameters related to mucositis, and investigating the impact of the intervention on the quality of life of patients. Methodology: This is a randomized, double-blind, parallel, single-center clinical trial to be conducted at the Borges da Costa Outpatient Clinic located at the Hospital das Clínicas of the Federal University of Minas Gerais in Belo Horizonte (HC-UFMG). Inclusion criteria involve adult patients, aged ≥ 18 years, of both sexes, diagnosed with colorectal cancer and candidates for first-line chemotherapy treatment with Capecitabine alone or in combination with Oxaliplatin, treated at HC/UFMG under the signature of the Informed Consent Form (ICF) and able to follow the research guidelines. The study was approved by the Research Ethics Committee of UFMG (CEP-UFMG) under protocol number CAAE 30177920.2.0000.5149. The study involves 80 participants distributed according to the chemotherapy protocol. Patients will be randomly divided into two groups designated as A and B: one control group receiving Maltodextrin, and the other intervention group receiving Symbiotic. The supplementation will be administered for 10 days, twice a day, before the start of chemotherapy treatment. Biological samples, such as feces and blood, will be collected for analysis of intestinal microbiota, short-chain fatty acid (SCFA) levels, presence of infection, intestinal permeability, and inflammatory markers. Biological collections will be performed at different time points throughout the study, including before supplementation (D0-D1), on the 10th day of supplementation (D10 pre-QTx), and on days 14 and 21 of the first chemotherapy cycle (D14-QTx and D21-QTx). Data will be collected through nutritional, anthropometric, and dietary assessments, including the Subjective Global Assessment (SGA), Anthropometric Assessment, Dietary Assessment (24h Recall and Food Frequency Questionnaire), as well as assessment of intestinal function and digestive complaints. Patients will be monitored daily, along with follow-up during treatment and data recording in the electronic medical record. Statistical analysis of the data will include sample size calculation, appropriate statistical tests, and an exploratory approach to evaluate clinical outcomes and study results. Expected Results It is expected that the results of this study will provide evidence on the efficacy of symbiotic supplementation in preventing oral mucositis in CRC patients undergoing chemotherapy. If the intervention proves to be effective, it could contribute to the development of more effective nutritional strategies in managing the side effects of oncological treatment, improving the quality of life and well-being of patients.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal tumor in the first oncological treatment
* Age over 18 years old
* Both sexes
* Eligible for protocol with capecitabine alone or associated with oxaliplatin
* Patients WITHOUT colostomy or WITH colostomy in the transverse/descending/sigmoid region
* Patient undergoing Radiotherapy treatment associated with Chemotherapy
* Patients residing in Belo Horizonte and the metropolitan region
* Patients who Accept and sign the Informed Consent Form (TCLE)

Exclusion Criteria:

* Diagnosis of gastrointestinal carcinoid and stromal tumor (GIST)
* Patients with Ileostomy
* Patients with colostomy in the ascending region of the colon
* Inflammatory bowel diseases: Crohn's and Colitis
* Use of antibiotics and antifungals in the last 15 days
* Use of prebiotic/probiotic and/or synbiotic in the last 15 days
* Use of antidiarrheal medication in the last 15 days
* Presence of fever and mucus discharge
* Pregnant or breastfeeding women
* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Intestinal Microbiota | six months after collecting data from all research participants
  Fecal calprotectin measured by ELISA.
Intestinal Microbiota | six months after collecting data from all research participants
  production of short-chain fatty acids.
Intestinal Microbiota | six months after collecting data from all research participants
  analysis of intestinal microbiota composition by sequencing the 16S rRNA gene.
Clinical Nutritional Diagnostic | six months after collecting data from all research participants
  Body mass index BMI in kg/m²
Nutritional Diagnostic | six months after collecting data from all research participants
  body weight in kg
Nutritional Diagnostic | six months after collecting data from all research participants
  height in m
Nutritional Diagnostic | six months after collecting data from all research participants
  circumferences in cm
Nutritional Diagnostic | six months after collecting data from all research participants
  body composition via triceps skin fold thickness in mm
Nutritional Diagnostic | six months after collecting data from all research participants
  hand grip resistance assessed by dynamometry in kg
Nutritional Diagnostic | six months after collecting data from all research participants
  Food Frequency Questionnaire
Nutritional Diagnostic | six months after collecting data from all research participants
  24-hour recall
Effect of the synbiotic in pain | six months after collecting data from all research participants
  Visual Analogue Score for Pain using the Visual Analogue Scale
inflammatory marker | six months after collecting data from all research participants
  Blood samples for Tumor Necrosis Factor TNF in pg/mL
inflammatory marker | six months after collecting data from all research participants
  Fatty Acid Binding Protein FABP2 in ng/mL
inflammatory marker | six months after collecting data from all research participants
  Lipopolysaccharide Binding Protein LBP in µg/mL
inflammatory marker | six months after collecting data from all research participants
  Lipopolysaccharide LPS in µg/mL
inflammatory marker | six months after collecting data from all research participants
  leukogram White Blood Cell Count in cells/µL
Questionnaire to assess quality of life | six months after collecting data from all research participants
  EORTC QLQ-C30 for all cancer patients
Questionnaire to assess quality of life | six months after collecting data from all research participants
  EORTC QLQ-CR29 for colorectal cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Simone de Vasconcelos Generoso, Principal Investigator — Escola de Enfermagem - UFMG
Locations (1):
- Escola de Enfermagem - UFMG, Belo Horizonte, Minas Gerais, Brazil